CLINICAL TRIAL: NCT01854203
Title: Combination of Cisplatin Plus Gemcitabine Induction Chemotherapy and Intensity-modulated Radiotherapy With or Without Concurrent Cisplatin for Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: Combination of Cisplatin Plus Gemcitabine Induction Chemotherapy and Intensity-modulated radiotherapyIntensity-modulated Radiotherapy With or Without Concurrent Cisplatin for NPC
Acronym: NPC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jian-jun Li, Dr, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ChiECRCT-2013003
Record Dates: First submitted 2013-05-10; First posted 2013-05-15 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Cisplatin; neoadjuvant chemotherapy; intensity-modulated radiation therapy; concurrent chemoradiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy, Intensity-Modulated; Gemcitabine; Cisplatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IInductive chemotherapy + concurrent cisplatin and IMRT (Experimental): Patients receive Gemcitabine (800mg/m2 on day 1,8) and cisplatin (80mg/m2 on day 1)of a 21 day cycle, patients received four cycles chemotherapy before the radiotherapy, then receive radical radiotherapy with IMRT and cisplatin (30 mg/m2，on day 1) repeated every weeks for 6 cycles during radiotherapy.
  Interventions: Drug: Inductive chemotherapy + concurrent cisplatin and IMRT
- Inductive chemotherapy + IMRT (Experimental): Patients receive Gemcitabine (800mg/m2 on day 1,8) and cisplatin (80mg/m2 on day 1)of a 21 day cycle, patients received four cycles chemotherapy before the radiotherapy, then receive radical radiotherapy with IMRT.
  Interventions: Drug: Inductive chemotherapy + IMRT

INTERVENTIONS:
Drug: Inductive chemotherapy + concurrent cisplatin and IMRT — Patients receive Gemcitabine (800mg/m2 on day 1,8) and cisplatin (80mg/m2 on day 1)of a 21 day cycle, patients received four cycles chemotherapy before the radiotherapy, then receive radical radiotherapy with IMRT and cisplatin (30mg/m2，on day 1) repeated every week for 6 cycles during radiotherapy.
  Other Names: Gemcitabine and cisplatin
  Arms: IInductive chemotherapy + concurrent cisplatin and IMRT
Drug: Inductive chemotherapy + IMRT — Patients receive Gemcitabine (800mg/m2 on day 1,8) and cisplatin (80mg/m2 on day 1)of a 21 day cycle, patients received four cycles chemotherapy before the radiotherapy, then receive radical radiotherapy with IMRT.
  Other Names: Gemcitabine and cisplatin
  Arms: Inductive chemotherapy + IMRT

SUMMARY:
Concurrent cisplatin-based chemotherapy plus radiotherapy increased the risk of treatment-related death and severe acute toxicity. The survival benefit of adding concurrent chemotherapy to intensity modulated radiation in patients with locoregionally advanced nasopharyngeal carcinoma is unclear. Gemcitabine plus cisplatin chemotherapy combine with radiotherapy was effective and well tolerated by patients with locoregionally advanced NPC.

DETAILED DESCRIPTION:
The purpose of this study is to compare gemcitabine plus cisplatin induction chemotherapy combine intensity-modulated radiotherapy with or without concurrent cisplatin in patients with locoregionally advanced nasopharyngeal carcinoma (NPC), in order to reevaluate the value of concurrent cisplatin when 4 cycles induction chemotherapy (gemcitabine+cisplatin) and IMRT is used.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing (according to World Health Organization (WHO 2005) histologically type).
* A Karnofsky performance status of at least 80;
* Tumor staged is according to the 7th American Joint Commission on Cancer edition as Stage III：T1-2N2M0, T3N0-2M0 Stage IVa：T4N0-2M0 Stage IVb：Any T、N3.
* Adequate marrow: a WBC ≥3.5×109 l-1; a platelet count ≥100×109 l-1; and hemoglobin levels ≥100 g/l.
* Normal liver function test: Alanine Aminotransferase (ALT)、Aspartate Aminotransferase (AST) <1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤2.5×ULN, and bilirubin ≤ULN.
* Adequate renal function: a creatinine clearance rate of at least 60 mL/min.
* Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

* WHO Type keratinizing squamous cell carcinoma.
* Age >65 years or <18 years.
* Distant metastasis,
* Treatment with palliative intent.
* Pregnancy or lactation.
* a history of previous radiotherapy in the nasopharyngeal region or previous chemotherapy.
* history of renal disease, unstable cardiac disease requiring treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3-year
  Overall survival is calculated from randomization to death from any cause.
Failure-free survival | 3-year
  Failure-free survival is calculated from the date of randomization to the date of the first failure at any site.
Locoregional failure-free survival | 3-year
  the latency to the first local failure
Distant failure-free survival | 3-year
  The latency to the first remote failure

SECONDARY OUTCOMES:
Difference in the complete response rates between the two treatment arms | 12 weeks after the completion of therapy

OTHER OUTCOMES:
Rates of toxicity | 3-years
  Rates of toxicity will also be compared. Rates will be compared by the chi-square test.The Chemotherapy toxicity include thrombocytopenia, leukocytopenia , anemia, granulocytopenia,damage to hepatic function, damage to renal function,constipation, diarrhea,vomiting and rash. The radiotherapy toxicities include mucositis, radiation dermatitis,dysphagia, xerostomia, skin fibrosis, trismus, hearing loss ane cranial neuropathy.

CONTACTS AND LOCATIONS:
Overall Officials: yong Su, M.D., Study Director — Sun Yat-sen University; Janjun Li, M.D., Principal Investigator — Sun Yat-sen University; Lizhi Liu, M.D., Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Cancer Center,Sun Yat-sen University, Guangzhou, Guangdong
  - State Key Laboratory of Oncology in South China, Cancer Center, Sun Yat-sen University, Guangzhou